CLINICAL TRIAL: NCT02601118
Title: Effects of Micro- and Subtle-expression Reading Skill Training in Medical Students
Brief Title: Micro-expression Reading Skill Training in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, M.D., Pusan National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: micro-expression reading
Record Dates: First submitted 2015-11-05; First posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- training group (Experimental): 41 training students were pre-tested before education with Micro Expression Training Tool (METT) and Subtle Expression Training Tool (SETT) at baseline and then, took second METT and SETT tests after a 1-hour class about interpreting micro and subtle expressions.
  Interventions: Other: Micro Expression Training Tool
- control group (No Intervention): 41 control students were pre-tested before education with METT and SETT at baseline and then, took the second tests without attend the training class.

INTERVENTIONS:
Other: Micro Expression Training Tool — The Micro Expression Training Tool (METT) and the Subtle Expression Training Tool (SETT) to help improve the non-verbal communication skills
  Arms: training group

SUMMARY:
This study was undertaken to investigate the effectiveness of the Micro Expression Training Tool (METT) and the Subtle Expression Training Tool (SETT) to help improve the non-verbal communication skills of medical students.

DETAILED DESCRIPTION:
Teaching and assessing communication skills is an important component of medical school curricula, and it is not easy for medical students to develop non-verbal communication skills without adequate training. This study was undertaken to investigate the effectiveness of the Micro Expression Training Tool (METT) and the Subtle Expression Training Tool (SETT) to help improve the non-verbal communication skills of medical students.

ELIGIBILITY:
Inclusion Criteria:

* Year 1 and 2 medical students, PNUSOM

Exclusion Criteria:

* incomplete survey response

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Expression Training Tool score | through study completion, 1 year
  difference of Micro and Subtle Expression Training Tool score between pre-test and post-test